CLINICAL TRIAL: NCT03357445
Title: Prospective, Multi Centre Evaluation of AVANTAGE® RELOAD Double Mobility Acetabular Cup - Clinical and Radiographic Outcomes
Brief Title: AVANTAGE® RELOAD Double Mobility Acetabular Cup -Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BMETEU.CR.EU49
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Primary Osteoarthritis; Post-Traumatic Arthritis; Inflammatory Joint Disease; Femoral Neck Fracture; Femoral Head Necrosis; Sequelae From Previous Hip Surgery; Osteotomies; Congenital Hip Dysplasia
Keywords: Total hip Arthroplasty; Hip implant
MeSH Terms: conditions — Femoral Neck Fractures; Hip Dislocation, Congenital

STUDY DESIGN:
Who Masked: Participant
Masking Description: The two subgroups will have the medical device with the following objectives:
  Subgroup 1 Prospective non Controlled to Document long term performance of AVANTAGE® RELOAD.
  Subgroup 2 Randomized Controlled Trial to Evaluate wear rate of E1 liner in comparison to ArCom® liner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgroup 1 (Other): Prospective non Controlled to Document long term performance of AVANTAGE® RELOAD
  Interventions: Other: Avantage Reload cup
- Subgroup 2 (Other): Randomized Controlled Trial to Evaluate wear rate of E1 liner in comparison to ArCom® liner
  Interventions: Other: Avantage Reload cup

INTERVENTIONS:
Other: Avantage Reload cup — Patients receiving the Avantage Reload acetabular cup in total hip arthroplasty

SUMMARY:
This is a Post Marketing Clinical Follow Up study (PMCF) on the AVANTAGE RELOAD dual mobility system cup.

DETAILED DESCRIPTION:
The study objective is to document the patients' survivorship at 10 years and evaluate the performances at 3 months, 1, 2, 3, 5, 7 and 10 years post-surgery of the AVANTAGE RELOAD cup. Secondary objective is to evaluate the polyethylene wear between E1 and ARCOM.

500 patients was the enrollment goal with 2 subgroups.

* Subgroup 1: prospective and non-controlled to satisfy ODEP (Orthopedic Device Evaluation Panel) requirements;
* Subgroup 2: randomized and controlled to compare the polyethylene wear between the Arcom and the E1 liners.

ELIGIBILITY:
Inclusion Criteria:

* Selection of subjects for this evaluation should be in accordance with the indications of the AVANTAGE® RELOAD with E1™ or ArCom™ liner specifically

  * Primary osteoarthritis
  * Post-Traumatic arthritis
  * Inflammatory joint disease (e.g. Rheumatoid arthritis)
  * Femoral neck fracture
  * Femoral head necrosis
  * Sequelae from previous hip surgery, osteotomies, etc.
  * Congenital hip dysplasia

Additional inclusion criteria include:

* Male or female
* 18 years of age or older
* Subjects willing to return for follow-up evaluations
* Subjects who read, understand study information and give written consent (specific local regulatory requirements)

Exclusion Criteria:

* Exclusion criteria should be in accordance with Contraindications for the AVANTAGE®

RELOAD:

Absolute contraindications include:

* Infection
* Sepsis
* Severe muscular, neurological or vascular deficiencies of the extremity involved
* Bone destruction or poor bone quality

Additional contraindications include:

* Subjects unable to co-operate with and complete the study
* Dementia and inability to understand and follow instructions
* Neurological conditions affecting movement
* Patient over 18 under law supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-10-14 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 years post-surgery
  Implant survivorship

SECONDARY OUTCOMES:
Harris hip scores | 10 years post-surgery
  To measure clinical efficacy
EQ-5D | 10 years post-surgery
  To measure clinical efficacy
Radiographic Evaluation | 10 years post-surgery
  Abnormalities determined on X-rays in the bone region surrounding the implant will be reported (radiolucencies, osteolysis, hypertrophy, subsidence, heterotopic ossification, etc)
Complications | 10 years post-surgery
  Eventual complications occurred including dislocations and revisions/removals

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (4):
- France (3):
  - CHU Cote de Nacre, Caen
  - Hôpital Renée Sabran, Giens
  - CHU Lapeyronie, Montpellier
- Hospital Novo Mesto, Novo Mesto, Slovenia